CLINICAL TRIAL: NCT05058963
Title: Virtual Mantram Repetition Program for Patients With Posttraumatic Stress Disorder and Substance Use Disorders
Brief Title: Virtual Mantram Program for Patients With PTSD and SUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 018/2019
Record Dates: First submitted 2021-07-13; First posted 2021-09-28 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2023-01

CONDITIONS: Post Traumatic Stress Disorder; Substance Use Disorders
Keywords: Post Traumatic Stress Disorder; PTSD; Trauma; Substance Use Disorder; SUD; Substance Abuse; Mantram; Group therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Substance-Related Disorders; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mantram repetition program (Experimental): Weekly 90 minute virtual group therapy sessions for 8 weeks run by two faciliators and will consist of 5-8 participants.
  Interventions: Behavioral: Mantram repetition program

INTERVENTIONS:
Behavioral: Mantram repetition program — Week 1: Define and describe the characteristics of a "mantram" as taught by Eknath Easwaran and how it relates to posttraumatic stress (PTSD) Week 2: Identify ways to choose and use mantram repetition for training attention and targeting craving.
  Introduction to substance craving and identify triggers for use. Week 3: Describe the relationship between the PTSD/stress response, mantram repetition and the "relaxation response" Week 4: Describe at least two benefits of slowing down versus automatic pilot for stress reduction Week 5: Describe at least two benefits of one-pointed attention versus multitasking for stress reduction Week 6: Demonstrate how one-pointed attention and slowing down complement each other for making healthy choices Week 7: List at least five strategies for making mantram repetition a part of your life Week 8: Discuss applications of mantram repetition, one-pointed attention and slowing down for overall health and substance use

SUMMARY:
The purpose of this study is to evaluate a virtual Mantram repetition program for adults with PTSD and substance use disorders. The program involves repetition of a personalized Mantram, which is a word or short phrase with spiritual meaning that is frequently repeated throughout the day. The program also involves slowing down thoughts and have one-pointed attention that help with stress.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate a virtual Mantram repetition program for adults with PTSD and substance use disorders. The program involves repetition of a personalized Mantram, which is a word or short phrase with spiritual meaning that is frequently repeated throughout the day. The program also involves slowing down thoughts and have one-pointed attention that help with stress.

The study starts with an eligibility and baseline assessment, which involves completing a series of questionnaires. Following these assessments, enrolled participants will be placed into a Mantram repetition program group led by two facilitators. This group will consist of 5 to 8 participants who will meet virtually every week for ninety minutes over an 8-week period. During this time, participants will also be asked to complete weekly self-reported questionnaires on their own. Additionally, at weeks 4 and 8, the participants will complete assessments and questionnaires with a member of the study team. The program will end after week 8. At week 12, participants will be invited to participate in a focus group to complete additional assessments, as well as be asked open-ended questions assessing the impact of the program on PTSD symptoms, substance use, and substance use cravings.

In summary, the Mantram group program will take 8 weeks to complete and the assessments will take approximately 12 weeks to complete. Participants will receive compensation of up to $200 for their participation.

ELIGIBILITY:
Inclusion Criteria:

* participants 18-years old or older
* fluent in English
* diagnosed with PTSD by a healthcare practitioner confirmed with the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5 past month version)
* diagnosed with past-year substance use disorder other than tobacco or caffeine by a healthcare practitioner confirmed by Structured clinical interview for DSM-5 (SCID-5)
* agreed not to participate in other therapies during the program (mindfulness, yoga, biofeedback, self-hypnosis or tai chi)
* willing to commit to attend all sessions

Exclusion Criteria:

* diagnosis of a severe or unstable medical illness that precludes safe participation in the study by a healthcare practitioner
* diagnosis of schizophrenia, schizoaffective disorder, or bipolar disorder; or current acute psychosis or mania by a healthcare practitioner
* participants with moderate or high risk of suicide upon screening by the Columbia Suicide Severity Rating Scale (C-SSRS)
* have an inability to communicate in English fluently enough to complete the questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Rate of retention in the group | 8 weeks
  Number of sessions completed for each participant, number of participants who withdraw and/or had non-attendance after enrollment in the study

SECONDARY OUTCOMES:
Alcohol consumption | 8 weeks
  Weekly alcohol consumption will be monitored using the timeline follow back interview
Drug consumption | 8 weeks
  Weekly drug consumption will be monitored using the timeline follow back interview
CAPS-5 PTSD Symptom Severity (past month) | Week 4, Week 8, Week 12 follow up
  Changes in PTSD symptoms and wellbeing will be monitored using the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) at the mid- and end-point of therapy and at follow up; 30-item questionnaire assessing 20 PTSD symptoms and overall PTSD severity; severity scale ranges from 0 to 4 with 0 = absence in symptoms to 4 being the highest symptom severity
Self-Rated PTSD Symptom Severity | 8 weeks
  Changes in PTSD symptoms severity will be monitored weekly using the PTSD Checklist for DSM-5 (PCL-5); 20-item checklist with scale from 0 to 4, where 0 means no endorsement and 4 means greatest level of PTSD-related distress.
Wellbeing | Baseline; Week 4; Week 8; Week 12 follow up. Scale Title: 12-item Short Form Health Survey , Minimum value: 0 , Maximum value : 100. The higher the score the better the outcome.
  Changes in wellbeing will be monitored at 3 time points using the 12-item Short Form Health Survey (SF-12)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Hassan, MD, MPH, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Ferkul S, Agabani Z, Minami O, Bormann J, Le Foll B, Lobo L, Hassan AN. The acceptability and feasibility of a virtual mantram program for patients with posttraumatic stress disorder and substance use disorders: mixed method results. BMC Complement Med Ther. 2024 Jan 2;24(1):9. doi: 10.1186/s12906-023-04312-1. PMID 38166894